CLINICAL TRIAL: NCT04484558
Title: Anxiety and Depression Disorder in Patient Treated With rTPA for Mangment of Acute Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ebtsam Tawfik, Principal investigator, Assiut University
Other Study IDs: 01001297992
Record Dates: First submitted 2020-02-16; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Acute Stroke; Anxiety Disorders; Depression
MeSH Terms: conditions — Stroke; Anxiety Disorders; Depression | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Actilyse — Infusion
  Other Names: rTpA

SUMMARY:
In fact theWorld Health Organization estimates that 2-3% in general populations of countries across the world tend to be affected by severe mental disorders (1) Thrombolytic therapy seems to be of great importance in achieving better quality of life in ischemic stroke patients who respond to this therapy(rTPA).

DETAILED DESCRIPTION:
There is a substantial body of evidenc suggesting a strong relation between neurotrophic factors and depression and anxiety pathogenesis (2,8) Brain-derived neurotrophic factor (BDNF), a member of the neurotrophic family known to regulate neuronal plasticity and survival , may play an important role in the pathophysiology of depression and anxiety (3,9).

Different studies indicated patients who were exposed to traumatic events have anxiety comorbidity and lower levels of serum BDNF compared to those without a history of traumatic events (4) .

BDNF has an antidepressant and anxiolytic effect which suggest that BDNF is implicated in the regulation of anxiety-related behaviors. which leads to a valine-to-methionine change in the proBDNF protein, was associated with lower activity-dependent secretion of BDNF (5)and has been implicated with increased susceptibility to neuropsychiatric disorders including depression, anxiety-related dysfunction, and bipolar disorder , all these studies suggest that BDNF is likely to be an important etiological factor in memory, depression and anxiety disorders (6,10).

BDNF arises from a precursor, proBDNF, which is cleaved to produce the mature protein through the tissue plasminogen activator (tPA) pathway, and represents one mechanism that can regulate the action of BDNFarises from a precursor, proBDNF, which is cleaved to produce the mature protein through the tissue plasminogen activator (tPA) pathway, and represents one mechanism that can regulate the action of BDNF (7).

The purpose of this study is to examine the quality of life after stroke of patients treated with thrombolysis .

ELIGIBILITY:
Inclusion Criteria:

1. age more than 40.
2. None of the pt had history of other psychiatric illness.
3. male and female.

Exclusion Criteria:

* 1-smoker. 2-substance abuser or dependence. 3-History of other psychiatric illness. 4-History of other neurological illness.

Ages: 40 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Data will be collected from the clinical interpretation of the patients at presentation and from the recent patients' medical records which have the full medical histories and examinations. All patients will be subjected to full neurological history and examination. The results of the above mentioned laboratory, investigations will be included in future analysis and interpretation of patients' abnormal neurological findings.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Detection and measureing anxiety and depressive symptoms in ischemic stroke patients treated with rtpA . | 15 minutes
  Hamilton depression and anxiety rating scale

SECONDARY OUTCOMES:
Measuring quality of life in patients with ischemic stroke treated wih rtpA . | 10 minutes
  Quality of life questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Musumeci G, Sciarretta C, Rodriguez-Moreno A, Al Banchaabouchi M, Negrete-Diaz V, Costanzi M, Berno V, Egorov AV, von Bohlen Und Halbach O, Cestari V, Delgado-Garcia JM, Minichiello L. TrkB modulates fear learning and amygdalar synaptic plasticity by specific docking sites. J Neurosci. 2009 Aug 12;29(32):10131-43. doi: 10.1523/JNEUROSCI.1707-09.2009. PMID 19675247
- [Background] Noble EE, Billington CJ, Kotz CM, Wang C. The lighter side of BDNF. Am J Physiol Regul Integr Comp Physiol. 2011 May;300(5):R1053-69. doi: 10.1152/ajpregu.00776.2010. Epub 2011 Feb 23. PMID 21346243
- [Background] Kauer-Sant'Anna M, Tramontina J, Andreazza AC, Cereser K, da Costa S, Santin A, Yatham LN, Kapczinski F. Traumatic life events in bipolar disorder: impact on BDNF levels and psychopathology. Bipolar Disord. 2007 Jun;9 Suppl 1:128-35. doi: 10.1111/j.1399-5618.2007.00478.x. PMID 17543031
- [Result] Li Y, Luikart BW, Birnbaum S, Chen J, Kwon CH, Kernie SG, Bassel-Duby R, Parada LF. TrkB regulates hippocampal neurogenesis and governs sensitivity to antidepressive treatment. Neuron. 2008 Aug 14;59(3):399-412. doi: 10.1016/j.neuron.2008.06.023. PMID 18701066